CLINICAL TRIAL: NCT04513184
Title: Randomized Clinical Trial of Intranasal Dexamethasone as an Adjuvant in Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edda Sciutto Conde (Other)
Collaborators: Hospital General de México Dr. Eduardo Liceaga (Other Government); Instituto Nacional de Cardiologia Ignacio Chavez (Other); El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Responsible Party: Sponsor-Investigator, Edda Sciutto Conde, Researcher, Universidad Nacional Autonoma de Mexico
Organization: Universidad Nacional Autonoma de Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DI/20/407/04/36
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Covid19
Keywords: Dexamethasone; SARS CoV-2 infection; COVID-19; Severe Acute Respiratory Syndrome; Nasal administration
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, controlled trial adult patients with confirmed COVID-19 infection
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard therapy (ST) only (Active Comparator): Control. Standard care and treatment only
  Interventions: Drug: IV Dexamethasone
- DXM (Experimental): Nasal dexamethasone plus Standard care and treatment
  Interventions: Drug: Nasal Dexamethasone

INTERVENTIONS:
Drug: IV Dexamethasone — 6 mg from Day 1 to 10 after randomization
  Other Names: ST
  Arms: Standard therapy (ST) only
Drug: Nasal Dexamethasone — 0.12 mg/kg/daily for 3 days from day 1, followed by 0.06 mg/kg/daily from day 4 to 10 after randomization.
  Other Names: Nasal DXM
  Arms: DXM

SUMMARY:
This Clinical Trial evaluates nasal administration of Dexamethasone as an adjuvant treatment strategy for non-critically ill hospitalized participants with SARS CoV-2 infection.

DETAILED DESCRIPTION:
Approximately 30% of the admitted patients with Covid-19 require admission to the intensive care unit for respiratory assistance, ranging from a high flow nasal cannula to invasive ventilation. These patients are affected by respiratory dysfunctions and even dysfunction of the brain respiratory control centers. Additionally, exacerbated inflammation leads to endothelial and coagulation disorders that aggravate the course of the illness. No effective therapy has yet been found to treat forms SARS-CoV-2 bass. One of the adjunctive therapeutic alternatives addressed is the use of intravenously administered glucocorticoids (GC), aimed at reducing exacerbated peripheral inflammation. They have been used at early stages of infection in high doses and with controversial results. In our laboratory at the Biomedical Research Institute from the National Autonomous University of Mexico (UNAM), we have shown that dexamethasone, a GC (DXM) administered intranasally, reaches the central nervous system through the olfactory nerve (alike various pathogens, including coronaviruses) and reduces neuroinflammation more effectively than when applied intravenously. Additionally, biodistribution studies indicate that the DXM is detectable from the first minute after its application, both in the central nervous system and in the respiratory system. The objective of this study is to evaluate the safety, efficacy and tolerability of dexamethasone in patients hospitalized with SARS-CoV-2 with moderate-severe forms, with an without the requirement of mechanic ventilation, including syndrome of acute respiratory distress or pneumonia (as diagnosed by CAT) with alveolar / interstitial lung involvement.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis of SARS-CoV-2 by real-time RT-PCR in oropharyngeal sample.
* 7 days or more after the start of the infection
* Hospitalized patients with moderate to severe respiratory complications that do not have received mechanical ventilation.
* Patients receiving standard therapy at the Hospital General de México Eduardo Liceaga.
* Signing of the informed consent form
* Patients of both sexes (non-pregnant female) 18 years of age or older will be eligible if they have a positive diagnostic sample by RT-PCR, pneumonia confirmed by chest imaging and oxygen saturation (SaO2) < 93% at ambient air or a ratio of the partial pressure of oxygen (PaO2) to the fraction of inspired oxygen (FiO2) (PaO2: FiO2) at 300 mg Hg or less

Exclusion Criteria:

* Patients participating in another research protocol.
* Patients receiving oral or intravenous glucocorticoids
* Immunosuppressed patients (including HIV infection)
* Glaucoma patients.
* Patients with allergy to dexamethasone.
* Pregnant or lactating women
* Concomitant autoimmune diseases
* Refusal by the patient or family to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Time of clinical improvement | 10 days after randomization
  Evaluation of the clinical status of patients after randomization, defined as a two point improvement in the WHO 7-point Ordinal Scale

SECONDARY OUTCOMES:
Time-to-death from all causes | 28 days after randomization
  All-cause mortality rates at 28 days after randomization
Time free from mechanical ventilation | 10 days after randomization
  Ventilator-free days, defined as alive and not requiring mechanical ventilation, at 10 days after randomization.
Viral load | 10 days after randomization
  Virological measurements, including proportions with detection of viral RNA over time and measurements of viral RNA titer area under the curve (AUC).
Length of hospital stay | 10 days after randomization
  Length of hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Edda Sciutto, PhD, Principal Investigator — Instituto de Investigaciones Biomédicas, UNAM
Locations (3):
- Mexico (3):
  - Hospital General de Mexico Dr. Eduardo Liceaga, Mexico City, Mexico City
  - Instituto Nacional de Cardiología Ignacio Chávez, Mexico City, Mexico City
  - El Instituto Nacional de Neurologia Y Neurocirugia Manuel Velasco Suarez, Mexico City, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Information exchange for research purposes
Supporting Information: Study Protocol, CSR
Time Frame: Upon study completion, by request

REFERENCES:
- [Derived] Cardenas G, Chavez-Canales M, Espinosa AM, Jordan-Rios A, Malagon DA, Murillo MFM, Araujo LVT, Campos RLB, Wong-Chew RM, Gonzalez LER, Cresencio KI, Velazquez EG, de la Cerda MR, Leyva Y, Hernandez-Ruiz J, Hernandez-Medel ML, Leon-Hernandez M, Quero KM, Moncivais AS, Diaz SH, Martinez IRZ, Martinez-Cuazitl A, Salazar INM, Sarmiento EB, Pena AF, Hernandez PS, Reynoso RIA, Reyes DM, Del Rio Ambriz LR, Bonilla RAA, Cruz J, Huerta L, Fierro NA, Hernandez M, Perez-Tapia M, Meneses G, Espindola-Arriaga E, Rosas G, Chinney A, Mendoza SR, Hernandez-Aceves JA, Cervantes-Torres J, Rodriguez AF, Alor RO, Francisco SO, Salazar EA, Besedovsky H, Romano MC, Bobes RJ, Jung H, Soldevila G, Lopez-Alvarenga J, Fragoso G, Laclette JP, Sciutto E. Intranasal dexamethasone: a new clinical trial for the control of inflammation and neuroinflammation in COVID-19 patients. Trials. 2022 Feb 14;23(1):148. doi: 10.1186/s13063-022-06075-5. PMID 35164840